CLINICAL TRIAL: NCT06456710
Title: Effect of Acceptance and Commitment Therapy on Stigma in College Students With Irritable Bowel Syndrome: a Randomized Controlled Study
Brief Title: Effect of a Psychological Intervention on Stigma: a Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yangzhou University (Other)
Responsible Party: Principal Investigator, Gao Yajun, Principal Investigator, Yangzhou University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YZUHL20220044
Record Dates: First submitted 2024-06-05; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Irritable Bowel Syndrome; Stigma; Psychological Intervention
Keywords: Irritable Bowel Syndrome; Stigma; Acceptance Commitment Therapy
MeSH Terms: conditions — Irritable Bowel Syndrome; Social Stigma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional IBS Health Education (Placebo Comparator): Patients were provided with IBS related knowledge (e.g., the pathogenesis of IBS and the reasons affecting the treatment effect), exercise guidance, drug guidance and dietary management precautions; and timely answers to patients' clinical problems and psychological support.
  Interventions: Behavioral: Conventional IBS Health Education
- Based on ACT Theory of Psychological Intervention (Experimental): A psychological intervention program based on ACT theory was implemented on top of the control group.
  Interventions: Behavioral: Based on ACT Theory of Psychological Intervention

INTERVENTIONS:
Behavioral: Conventional IBS Health Education — Patients were provided with IBS related knowledge (e.g., the pathogenesis of IBS and the reasons affecting the treatment effect), exercise guidance, drug guidance and dietary management precautions; and timely answers to patients' clinical problems and psychological support.
  Arms: Conventional IBS Health Education
Behavioral: Based on ACT Theory of Psychological Intervention — On the basis of the control group, the stigma intervention program of college students with IBS based on ACT theory was implemented. The duration of intervention was 40 to 50 minutes for 6 times, once a week for 6 weeks.
  Week1: established relationships; introduced the core contents of ACT, the treatment process, and the effects of application.
  Week2: encouraged to express negative emotions and behaviors; made patients accept the disease.
  Week3: explained the importance of coping with negative emotions; instructed to separate negative thoughts from reality through cognitive dissociation exercises.
  Week4: changed the concept of "self" and actively accepted IBS; guided to focus on the current life and true self.
  Week5: introduced the values in ACT; helped clarify the values; guided to build confidence and focused on the core values.
  Week6: introduced the importance of commitment to action; developed goals and plans together; encouraged to strengthen the use of ACT.
  Arms: Based on ACT Theory of Psychological Intervention

SUMMARY:
The purpose of this study was to construct a Stigma intervention program for college students with Irritable Bowel Syndrome (IBS) based on the Acceptance and Commitment Therapy (ACT) theory and to investigate the effectiveness in reducing stigma in IBS patients with the aim of enhancing their mental health and improving their quality of life.

DETAILED DESCRIPTION:
Using purposive sampling method, 84 college students with irritable bowel syndrome (IBS) accompanied by a sense of shame who met the inclusion and exclusion criteria from June 2023 to January 2024 in a comprehensive university in Yangzhou City were selected for the study. Using the method of random grouping, the patients who met the inclusion and exclusion criteria were numbered and randomly divided into the control group and the intervention group by computer random number procedure. Because individual patients fell out during the study, the final sample size for inclusion in the study was 80 cases, with 40 cases in each group. The control group was given conventional health education on irritable bowel syndrome, and the intervention group was given a 6-week acceptance and commitment therapy-based intervention programme for college students with irritable bowel syndrome based on stigma, with a 6-week intervention period and a 3-month follow-up period. The ANOVA of repeated measures data was used to analyse the trends in the Stigma, Psychological flexibility (PF), Self-acceptance (SA) and Quality of Life (QOL) score trends over time to assess the effects of the intervention. A single-blind method was used in this study, and only the outcomes assessor was blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patients with IBS who meet the Rome IV diagnostic criteria;
* Duration of IBS disease≥0.5 years;
* The Perceived Stigma Scale in IBS (PSS-IBS) total score≥80;
* Patients can proficiently use WeChat and participate in remote follow-ups;
* Understand the research content, participate voluntarily and sign the informed consent.

Exclusion Criteria:

* Patients with other intestinal diseases or serious primary diseases;
* Patients with comorbid psychiatric diseases;
* Patients who engaged in psychological workers or received psychological counseling within 3 months;
* Patients who have recently participated in or are currently participating in other similar studies.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Stigma | Baseline, 1 and 3 months post-intervention
  The Perceived Stigma Scale in IBS (PSS-IBS) was used to assess perceived stigma in terms of disease disclosure, attitude and knowledge about disease, disease efficacy, severity, and blame. The scale has 10 entries with 6 dimensions and is scored on a 5-point Likert scale from 0 to 4, with total scores ranging from 0 to 240, with the higher scores indicating the higher the level of perceived stigma. A score of 1 to 80 indicates mild, a score of 81 to 161 is moderate, and a score of > 161 is severe.

SECONDARY OUTCOMES:
Psychological flexibility (PF) | Baseline, 1 and 3 months post-intervention
  Acceptance and Action Questionnaire-II (AAQ-II) was used to assess the patients' level of psychological flexibility. The scale consists of 7 entries and is scored on a 7-point Likert scale from 1 to 7, with total scores ranging from 7 to 49. The higher the score, the lower the psychological flexibility, the higher the degree of empirical avoidance.
Self-acceptance (SA) | Baseline, 1 and 3 months post-intervention
  Self-Acceptance Questionnaire (SAQ) consists of two dimensions (self-acceptance and self-evaluation) with a total of 16 entries. The scale is scored on a 4-point Likert scale from 1 to 4, with total scores ranging from 16 to 64. A higher score indicates a higher level of self-acceptance.
Quality of Life (QOL) | Baseline, 1 and 3 months post-intervention
  IBS quality of life (IBS-QOL) consisted of 34 items with 8 dimensions, namely, anxiety, behavior disorder, body ideation, health worry, food avoidance, social function, sexual behavior, and interpersonal relationship. The scale adopts Likert's 5-point scale, with scores ranging from 1-5 from the lowest to the highest. The score of each dimension is converted by the formula to make the value range from 0 to 100. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Yajun Gao, Master, Principal Investigator — Yangzhou University
Locations (1):
- Yangzhou University, Yangzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
No plans to provide IPD

REFERENCES:
- [Result] Dear BF, Scott AJ, Fogliati R, Gandy M, Karin E, Dudeney J, Nielssen O, McDonald S, Heriseanu AI, Bisby MA, Sharpe L, Jones MP, Ali S, Titov N. The Chronic Conditions Course: A Randomised Controlled Trial of an Internet-Delivered Transdiagnostic Psychological Intervention for People with Chronic Health Conditions. Psychother Psychosom. 2022;91(4):265-276. doi: 10.1159/000522530. Epub 2022 Apr 1. PMID 35367986

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT06456710/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT06456710/ICF_001.pdf